CLINICAL TRIAL: NCT02455219
Title: Investigating the Use of Siemens Prototype UHRSZ Collimator for Imaging DatScan SPECT/CT Imaging
Brief Title: DatScan With Prototype Collimator
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 201503M65881
Record Dates: First submitted 2015-05-15; First posted 2015-05-27 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Prototype UHRSZ (UltraHigh Resolution Smart Zoom) Collimator — In DATScan SPECT scans, the UHRSZ collimator will be exchanged for the standard collimator following completion of the clinically ordered scan. A scanning sequence will be repeated with the prototype collimator in place. Images from the two scanning sequences will be compared.

SUMMARY:
A collimator is an accessory to a SPECT/CT scanner. It can be compared to a camera lens or filter that enhances or improves photos. The prototype collimators are able to magnify target organs about four times compared to the current collimators. In this study we are validating a new collimator design, which will allow for quantitative measurement of dopamine receptors within the brain, not previously performed using a single photon gamma camera.

DETAILED DESCRIPTION:
Previously PET/CT has been used for this measurement but the L-DOPA is not FDA approved and thus of limited availability. DatScan (I123 ioflupane) is an FDA approved and clinically indicated biomarker, which has a high binding affinity for presynaptic dopamine transporters (DAT) in the brains of mammals, in particular the striatal region of the brain. A feature of Parkinson's disease is a marked reduction in dopaminergic neurons in the striatal region. By introducing an agent that binds to the dopamine transporters a quantitative measure and spatial distribution of the transporters can be obtained. The use of SPECT/CT (with the new validated collimators) and the FDA approved DATScan biomarker would allow for readily available diagnosis of Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* all patients referred

Exclusion Criteria:

* anyone who wishes to not participate and cannot lay on the table for an additional 30 minutes.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to Nuclear Medicine for a clinically indicated DatScan for the diagnosis of Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
comparing images with prototype collimator to clinical images | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States